CLINICAL TRIAL: NCT00176995
Title: Phase II, Open-Label Study of the Effect of 15% Eflornithine Hydrochloride Cream on Facial Hair of Men of African-American Descent With Pseudofolliculitis Barbae: A Laser Scanning Confocal Microscopy and Video Imaging Study
Brief Title: Effect of 15% Eflornithine Hydrochloride Cream on African-American Males With Pseudofolliculitis Barbae
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hordinsky, Maria K., MD (Individual)
Organization: University of Minnesota (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 9902M00119
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-11-13 (Estimated); Status verified 2006-11

CONDITIONS: Pseudofolliculitis Barbae
MeSH Terms: conditions — pseudofolliculitis barbae

INTERVENTIONS:
Drug: 15% Eflornithine Hdyrochloride

SUMMARY:
This trial is designed to gain insight into the mechanism of action of eflornithine hydrochloride in men and to aid in determining if this compound is deserving of further development for a pseudofolliculitis barbae indication. This study will also provide knowledge which will be useful in designing future PFB trials in this indication is pursued.

DETAILED DESCRIPTION:
The proposed mechanism of action of eflornithine hydrochloride for treatment of hair growth is that it reduces the rate of cell growth within the hair follicle by inhibition of the enzyme ornithine decarboxylase (ODC). In preclinical studies eflornithine hydrochloride was shown to inhibit ODC and decrease hair mass. In sheep, systemic inhibition of ODC by eflornithine hydrochloride markedly altered not only the length and diameter of hair fibers, but also the portion of the hair fiber cross-section occupied by paracortical cells, which are primarily found in straight hairs. In a Phase II study evaluating the effect of the drug in the treatment of female hirsutism, it was anecdotally noted that those who also had PFB showed an improvement in this condition.

ELIGIBILITY:
Inclusion Criteria:

* Males age 18 or older of African American descent.
* History of PFB localized to the beard area of at least 2 years duration confirmed by a dermatologist.
* PFB grade 3 (ingrown hairs and 20 or more papules of 2mm or greater in diameter with inflammation with minimal pustules) or greater involving the beard area of the face.
* Customary frequency of removal of facial hair by wet shaving at least once per week.

Exclusion Criteria:

* Use of topical medications on the face within 2 weeks prior to treatment.
* Use of systemic steroids, antibiotics, lithium or isotretinoin within 2 months prior to pretreatment. Use of etretinate or acitretin within one year prior to pretreatment.
* Use of systemic antiandrogens, spironolactone, growth hormone, immunostimulants. immunosuppressants, 5-alpha reductase inhibitors. minoxidil dehydroepiandrosterone (DHEA) or other medications considered to have an effect on hair growth within 6 months prior to pretreatment.
* Use of physical hair removal techniques (laser, electrolysis, epilation) or chemical removal products (depilatories, waxing, sugaring) within 4 weeks prior to pretreatment.
* Presence of bacterial infections in the beard area including abscesses (3 or more) covering greater than 10% of the face and/or severe inflammatory acne.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 1999-03; Study Completion 2000-10

PRIMARY OUTCOMES:
Observation of changes in actin filament/stress fibers orientation formation and location in the beard hair follicles in African American men before and after treatment.

SECONDARY OUTCOMES:
Observation of changes in binding of this lectin or orthocortical cells of beard hair follicles in African American men before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, MD, Principal Investigator — University of Minnesota; Marna Ericson, Ph D, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States